CLINICAL TRIAL: NCT04472988
Title: The Effects of Eye Movement Desensitization and Reprocessing on Autoimmune Thyroiditis in Adults: a Randomized Controlled Trial
Brief Title: Eye Movement Desensitization and Reprocessing on Autoimmune Thyroiditis in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Maria Magdalena Macarenco, The effects of Eye Movement Desensitization and Reprocessing on Autoimmune Thyroiditis in adults: a randomized controlled trial, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 39/27.02.2019
Record Dates: First submitted 2020-07-07; First posted 2020-07-16 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hashimoto
Keywords: Hashimoto; Autoimmune thyroiditis; Eye Movement Desensitization adn Reprocessing; Trauma
MeSH Terms: conditions — Hashimoto Disease; Thyroiditis, Autoimmune; Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: During the study an endocrinologist who will be blinded to randomization groups will evaluate the biological markers of the participants at baseline, post-treatment and follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eye Movement Desensitization and Reprocessing (Experimental): 30 participants will be randomly allocated to the EMDR group. They will receive a 90 minutes session of EMDR each week for twelve weeks. The sessions will be conducted by clinicians or psychotherapists specialized in EMDR, and the participants will be randomly allocated to them.
  EMDR is a structured, goal-oriented, short-term intervention organized around traumatic or stressful memories. This method was discovered in 1981 by F. Shapiro and represented an evidence-based treatment, one of the two first-line trauma treatment recommended for use with adults (NICE, 2005; World Health Organization, 2013). EMDR proved effective by hundreds of researches and has also been shown to be useful in alleviating physical symptoms such as pain or increased autonomic activity. But to our knowledge, research on EMDR efficacy in the treatment of autoimmune thyroiditis has not been previously reported.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing
- Placebo (Placebo Comparator): 30 participants will be randomized to the placebo group. The placebo goup will receive an intervention that does not include working on past traumatic memories, it will be more focused on present and future.
  Interventions: Other: Placebo
- Treatment as Usual (Active Comparator): 30 participants will be randomized to this group. They will continue only the medical treatment for Hashimoto their doctor prescribed to them.
  Interventions: Drug: Treatment as Usual

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing — The first session will be assigned to the assessment and the exploration of the personal history and for presenting the method to the client. Then, each case will be conceptualized according to the Model of Two Method Approach and the protocol for the treatment will be used. The procedure will be organized around targeting the most ten disturbing memories which happened before the illness debut, including stressful or traumatic memories from childhood. The rationale behind this approach is that adverse events leave traces in the neural network of an individual in such a way that these cause a variety of emotional or cognitive symptoms. If we consider the illness as being also a "symptom" of a traumatic past, then we expect that by accessing the dysfunctionally stored memory and stimulating the innate processing system, the symptoms of the illness diminish.
  Arms: Eye Movement Desensitization and Reprocessing
Other: Placebo — The participants randomised in this group will receive a protocol focused only on present and future (present symptoms, daily problems, future projects). The psychologist will lead the discussion anywhere except for the past.
  Arms: Placebo
Drug: Treatment as Usual — The participants randomised in this group will continue taking the classical treatment prescribed for Hashimoto (Levothyroxine)
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to evaluate whether Eye Movement Desensitization and Reprocessing (EMDR) is effective in decreasing the level of autoantibodies of patients with autoimmune thyroiditis. The investigators hypothesize that processing traumatic memories from events that happened before the illness onset will have a positive impact first on the psyche (a) by decreasing the level of dissociation, alexithymia, anger, and (b) by increasing the quality of life and emotional regulation, than those in the control group. Secondly, it will have an impact on the biological level, by decreasing the level of autoantibodies, antithyroglobulin antibody (anti-Tg) and anti-thyroid peroxidase antibody (anti-TPO), which are the main antibodies detected in chronic autoimmune thyroiditis.

DETAILED DESCRIPTION:
Hashimoto thyroiditis is an autoimmune disease that leads to chronic inflammation of the thyroid gland. This is considered the most common autoimmune disorder, and the most common endocrine disorder. Psychological trauma has been suggested as a possible factor in the pathogenesis and development of autoimmune diseases. Although a diversity of psychotherapeutic interventions have been studied in adults with autoimmune diseases, there is a lack of psychological research and randomized controlled trials in the field of the Hashimoto disease.

This study is designed to be a clinical trial with three arms: one experimental and two control groups. The experimental group receives EMDR, one control group receive placebo and the other is a waiting list. 90 out-patients with Hashimoto disease will be randomly assigned to the three groups. The investigators hypothesize that the therapeutic gains will be more significant in the experimental condition than in the control groups at the completion of the therapy and that this will be maintained at the 3-month follow-up.The EMDR group undergoes a 90 minutes session of EMDR each week for twelve weeks.The sessions will be conducted by clinicians or psychotherapists specialized in EMDR. The placebo group will receive a similar amount of time of placebo intervention. If therapy is efficient on the autoimmune disorder, participants in the control groups will be reallocated to EMDR after the experimental treatment will come to an end.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-55 years;
* confirmed autoimmune thyroiditis diagnosis
* at least one biological marker Anti-thyroid peroxidase (anti-TPO) antibodies or thyroglobulin antibodies (TgAb) exceeds the reference range

Exclusion Criteria:

* the presence of psychotic symptoms
* currently receiving another form of psychological treatment;
* under psychotropic medication;
* neurodevelopmental disorders (intellectual disability, communication disorders, autism spectrum disorders, ADHD);
* neurocognitive disorders;
* substance abuse;
* serious legal or health issues that would prevent from regularly attending
* patients with autoimmune thyroiditis with biological markers within the reference range

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Measurement of anti-thyroid peroxidase levels (anti-TPO) | baseline to 6 months
  Measurement of anti-thyroid peroxidase in adults with Hashimoto at baseline, post-treatment and follow-up, after trauma therapy with EMDR
Measurement of thyroglobulin levels (TgAb) | baseline to 6 months
  Measurement of thyroglobulin antibodies levels in adults with Hashimoto at baseline, post-treatment and follow-up, after trauma therapy with EMDR

SECONDARY OUTCOMES:
State-Trait Anger Expression Inventory | Baseline to 6 months
  Perceptions about anger expression in adults with Hashimoto will be measured at baseline, post-treatment and follow-up, after EMDR treatment. The inventory assesses a various area of anger and the traits of experiencing anger. Participants are asked to respond to 44 items using a 4-point scale ("Not at all" to "Almost always").
Toronto Alexithymia Scale | Baseline to 6 months
  Perceptions about alexithymia will be measured at baseline, post-treatment and follow-up, after EMDR treatment. Toronto Alexithymia Scale is a 20 item self-report instrument, with each item rated on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree).
Dissociative Experiences Scale | Baseline to 6 months
  Perceptions about the levels of dissociation will be measured at baseline, post-treatment and follow-up, after EMDR treatment. The instrument is a self-assessment questionnaire used to screen for dissociative symptoms. It consists of 28 items that assess the frequency and severity of a wide range of dissociative experiences using an eleven-point visual analog scale (0%-100%).
The Depression Anxiety Stress Scales | Baseline to 6 months
  Perceptions about depression, anxiety and stress levels will be measured at baseline, post-treatment and follow-up, after EMDR treatment. The instrument is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three scales contains seven items.
The World Health Organization Quality of Life | Baseline to 6 months
  Perceptions about the quality of life will be measured at baseline, post-treatment and follow-up, after EMDR treatment. The instrument is a 26-item self-report tapping into the following broad domains: physical health, psychological health, social relationships, and environment.

OTHER OUTCOMES:
The Difficulties in Emotion Regulation Scale | Baseline to 6 months
  Perceptions of the emotion regulation will be measured at baseline, post-treatment and follow-up, after EMDR treatment. The instrument is designed to assess clinically relevant difficulties in emotion regulation.
The Outcome Rating Scale and Session Rating scale | Baseline to 6 months
  This scales are very brief and feasible measures for tracking client well-being and the quality of the therapeutic alliance. The Outcome Rating Scale will be completed by the participant at the beginning of each of the 12 sessions. The Session Rating Scale will be completed by the participant at the end of each of the 12 sessions.
Intent-to-Attend Scale | Baseline to 6 months
  The scale is a single-item measure. Participants rate their intention on a nine-point Likert scale, at the end of each session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bucharest, Bucharest, Romania